CLINICAL TRIAL: NCT07000526
Title: Inhaled Sedation in Critically Ill Patients: a Multicentre Randomized Clinical Trial
Brief Title: Inhaled Sedation in Critically Ill Patients
Acronym: IS-CRITIC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, José Manuel Añón, Head of Department of Critical Care Medicine, Instituto de Investigación Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP6844; 2024-518521-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sedation; Airway Extubation
Keywords: Inhaled sedation; Mechanical ventilation; Delirium
MeSH Terms: conditions — Delirium | interventions — Isoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Inhaled sedation with Isoflurane. Initial dose: 3 mL/h. Gradual dose increase until target RASS is achieved. Do not exceed 14 mL/h. Guided by end tidal isoflurane concentration (EtISO), the recommended maximum dose for prolonged use is 1%. Short periods at up to 1.5% may be considered. If the target RASS is not achieved at the maximum dose, a second hypnotic agent may be added.
  Interventions: Drug: Isoflurane
- Control group (Active Comparator): Intravenous sedation with propofol (20 mg/mL). Initial dose: 0.5-1 mg/kg/h. Gradual dose increase until target RASS is achieved. Do not exceed 4 mg/kg/h. If the target RASS is not achieved at the maximum dose, a second hypnotic agent may be added.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Isoflurane — Inhaled sedation with isoflurane via Sedaconda ACD-S
  Other Names: Inhaled sedation with Isoflurane
  Arms: Study group
Drug: Propofol — Intravenous sedation with Propofol 20 mg/ml
  Other Names: Intravenous sedation with Propofol
  Arms: Control group

SUMMARY:
The proposal of this study is to compare inhaled sedation with isoflurane administered via the Sedaconda ACD-S system with intravenous sedation with propofol. Patients will be randomized 1:1 to receive either inhaled sedation with isoflurane administered via the Sedaconda ACD device (Sedana Medical, Uppsala, Sweden) or intravenous propofol. The primary endpoint is the number of ventilator-free days at 28 days after randomization.

DETAILED DESCRIPTION:
Justification: Isoflurane has recently emerged as an attractive alternative for intensive care unit (ICU) sedation. Due to their favorable pharmaco-kinetic and dynamic profile, this agent has been progressively introduced into clinical practice. Isoflurane has proven to be non-inferior to propofol in terms of efficacy and safety and it has been suggested that it may facilitate ventilator weaning. However, no differences in length of mechanical ventilation were found. These studies have focused on short sedation durations. In fact, long-term effects and outcomes associated with isoflurane for ICU sedation are not yet fully understood.

Hypothesis: Inhaled sedation with isoflurane administered via the Sedaconda ACD-S system in critically ill patients leads to a shorter duration of mechanical ventilation at 28 days and a reduced length of ICU stay compared to intravenous sedation with propofol.

Main objective: To compare the number of ventilator-free days at day 28 post-randomization between critically ill patients receiving sedation with isoflurane versus those receiving intravenous sedation with propofol in critically ill patients expected to require more than 48 hours of invasive mechanical ventilation. Key secondary objective: To compare the number of ICU-free days at day 28 post-randomization in both treatment arms. Secondary objectives: To compare time to extubation after sedation withdrawal, efficacy in maintaining a target level of sedation, compare the percentage of patients requiring one or more additional hypnotics, compare the incidence and duration of delirium at day 28, assess mental, cognitive, and quality of life status at 90 days post-hospital discharge between both treatment groups.

Methodology: Phase IV, low-intervention, open-label, multicenter, randomized controlled trial with intention-to-treat analysis including mechanically ventilated patients expected to require a minimum of 48 hours of mechanical ventilation with a RASS score between -3 and -5. Patients will be randomized 1:1 to receive inhaled sedation with isoflurane administered via the Sedaconda ACD device (Sedana Medical, Uppsala, Sweden) or intravenous sedation with propofol. A total of 620 patients will be included from a pool of 22 participating centers.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients receiving mechanical ventilation, with an anticipated duration >48 hours after randomization, and requiring deep sedation (target RASS between -3 and -5).

Exclusion Criteria:

* Contraindication to isoflurane or propofol
* Allergy to isoflurane or propofol
* Cardiopulmonary arrest
* History of ventricular tachycardia or long QT syndrome
* Tidal volume < 300 mL or PaCO₂ > 50 mmHg at the time of randomization.
* Invasive mechanical ventilation for more than 48 hours at the time of randomization.
* Pregnancy
* Breast feeding
* Acute neurological condition
* ECMO
* ECCO2R
* Active humidification strictly required
* Burns
* Lack of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days at day 28 from randomization | From randomization until day 28
  Number of days between randomization and day 28 during which the patient is alive and free from invasive mechanical ventilation. Patients who die before day 28, or who remain on mechanical ventilation at day 28, are assigned zero ventilator-free days.

SECONDARY OUTCOMES:
Key secondary objective: ICU-free days at day 28 post-randomization | From randomization until day 28
  Number of days between randomization and day 28 during which the patient is alive and free from the ICU. Patients who die before day 28, or remain in the ICU on day 28, are assigned zero ICU-free days.
Time to extubation | From randomization until day 28
  Mean number of hours from sedation withdrawal to successful extubation.
Administration of rescue sedation | From randomization until day 28
  Number of patients requiring the addition of one or more hypnotics
Sedation efficacy | From randomization until extubation or day 28
  Difference between the target sedation level and the actual measured level using Richmond Agitation Sedation Scale (RASS). Possible RASS score ranges from -5 (unarousable) to +4 (combative)
Number of Participants With Delirium | From randomization until extubation or day 28
  Number of patients with delirium using the Confusion Assessment Method in ICU (CAM-ICU)
Mortality | From randomization to day 60
  All cause mortality at 60 days from randomization
Number of Participants With Psychological disorders | at 90 days of hospital discharge
  Psychological status assessed using: 1.- Hospital Anxiety and Depression Scale (HADS). score of 8 or greater on the anxiety or depression subscale is used to identify symptoms of clinically significant anxiety or depression. 2.- Impact of Event Scale - Revised (IES-R), a self-report measure designed to assess the severity of post-traumatic stress disorder. Optimal screening threshold established as 1.6 (Consensus Conference on Prediction and Identification of Long-Term Impairments After Critical Illness. Crit Care Med 2020)
Number of Participants With Cognitive Disorders | at 90 days of hospital discharge
  Cognitive status assessed using Montreal Cognitive Assessment (MoCA) test. Total score ranges from zero to 30. Mild cognitive impairment: 18-25, moderate: 10-17, and severe: less than 10 (Consensus Conference on Prediction and Identification of Long-Term Impairments After Critical Illness. Crit Care Med 2020)
Number of Participants With Treatment-Related Adverse Events | From randomization to day 28
  Number of participants who experience at least one adverse event of special interest, deemed by the investigators to be related to the administered hypnotic, including events of mild, moderate, severe intensity, as well as serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: José M. Añón, MD, PhD, Principal Investigator — Hospital Universitario La Paz. IdiPAZ
Locations (22):
- Spain (22):
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital Universitario Doctor José Molina Orosa, Arrecife, Lanzarote-Canary Islands
  - Hospital Universitario de Albacete, Albacete
  - Hospital Germans Trias i Pujol, Badalona
  - Corporacio Sanitaria Parc Taulí, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Valle de Hebron, Barcelona
  - Hospital General Universitario Santa Lucía, Cartagena
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario La Paz, Madrid
  - Hospital Univeritario Puerta de Hierro, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid
  - Hospital Reina Sofía, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Joan XXIII, Tarragona
  - Hospital Universitario de Toledo, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Rio Hortega, Valladolid

IPD SHARING:
Plan to Share IPD: No